CLINICAL TRIAL: NCT05408507
Title: Feasibility and Acceptability of the ABC123 Framework for Advanced Cancer Care
Brief Title: Care Planning Framework in Advanced Cancer (ABC123)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-5030.cc; NCI-2022-01951 (Other: CTRP); 25A9726 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2022-05-17; First posted 2022-06-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Cancer
Keywords: incurable cancer; geriatric oncology; goals of care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older patients with advanced cancer (Experimental): Patients over 60 years old with advanced, incurable cancer.
  Interventions: Behavioral: ABC123 Framework

INTERVENTIONS:
Behavioral: ABC123 Framework — This care planning framework aims to implement existing tools in geriatric medicine, palliative medicine, and medical oncology to aid in cancer care planning for older adults with newly diagnosed incurable advanced cancer and to test the delivery of goal-concordant care. This patient-centered intervention is the ABC123 care planning framework in parallel with usual care that includes a physical function assessment, chemotherapy toxicity estimate calculation, and a guided goals of care discussion.

SUMMARY:
Pilot study assessing the feasibility and acceptability of the ABC123 framework, as well as goal concordance between patient and clinician stated goals. Patients >60 years old with recently diagnosed advanced, incurable cancer in for a first consultation at a participating medical oncology clinic. The team will pilot test the ABC123 framework delivery by an advanced practice provider working with a medical oncologist to inform the overall care planning process. This framework will routinely incorporate and implement existing resources from these 3 transdisciplinary tenets (geriatric, oncology, and palliative medicine) into initial care planning in a patient-centered manner. The team will follow patients from initial care planning to 6 months post-intervention and assess additional stakeholder feedback on barriers and facilitators to implementation.

DETAILED DESCRIPTION:
The ABC123 care planning framework is aimed at increasing care alignment delivered to older patients with advanced cancer by combining existing tools that represent the principles of geriatrics, oncology, and palliative care. In this pilot study, our primary goals are to assess the feasibility and acceptability of the ABC123 care planning framework and evaluate the framework's impact on the provision of care that aligns with the goals and values of patients. Participants will participate in a series of visits and follow-ups meant to implement and evaluate the ABC123 care planning framework that will take place over the course of six months. The first two visits will consist of 1) a short physical performance battery (SPPB) and estimation of potential for grade 3 chemotherapy toxicity using the Cancer and Aging Research Group chemotherapy toxicity calculator and 2) guided goals of care discussion with an Advanced Practice Provider based on the findings from visit 1. During 1, 3, and 6-month follow-up sessions, participants will complete a survey consisting of several commonly used questionnaires and an interview about experiences and goals. Care providers and institutional stakeholders will also be interviewed at 1, 2, and 3 years after initial implementation to understand experiences and assess the feasibility if the ABC123 framework.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Age >65 years old, or >60 with at least one deficit on a geriatric screen.
3. Stated willingness to comply with all study procedures and be available for the duration of the study
4. Diagnosis of a solid-tumor cancer that is not curable with surgery or radiation within the 6 mos. prior to consenting. And that would potentially be treated with systemic cytotoxic chemotherapy. If molecular marker status is pending for a particular tumor, patients may still be approached for enrollment in the study.
5. New patient consultation within the UCHealth Denver Metro system or newly diagnosed with recurrent metastatic/incurable disease
6. English speaking only for the pilot portion

Exclusion Criteria:

1. Have a diagnosis of a different advanced cancer that has required systemic therapy
2. Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility measured through recruitment | 3 years
  Recruitment (proportion of those approached who actually enroll)
Feasibility measured through retention in sessions | baseline to visit 2
  Retention number of those completing both clinic sessions
Feasibility measured through retention in follow up | baseline to 6 month follow up
  Retention number of those completing both sessions, and follow up

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kessler, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No